CLINICAL TRIAL: NCT03237208
Title: Patients Undergoing Routine Transcutaneous Electrical Nerve Stimulation Treatment in Patients With Renal Colic Who Admitted to the Emergency Department: A Randomized Double Blind Placebo-controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation Treatment of Renal Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08.06.2017/02
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Renal Colic
Keywords: Transcutaneous electrical nerve stimulation; emergency medicine
MeSH Terms: conditions — Renal Colic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Active Comparator): Patients receiving the real transcutaneous electrical nerve stimulation (TENS) with 100 hertz, pulse width 200 microseconds, voltage 2 milliampere
  Interventions: Device: TENS
- placebo group (Sham Comparator): Patients receiving the application of transcutaneous electrical nerve stimulation, but transcutaneous electrical nerve stimulation will not be activated.
  Interventions: Device: placebo group

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation (TENS) treatment will be activated.
  Arms: TENS
Device: placebo group — Transcutaneous electrical nerve stimulation treatment will not be activated.
  Arms: placebo group

SUMMARY:
The aim of the present trial was to investigate the analgesic efficacy and safety of Transcutaneous electrical nerve stimulation treatment in patients with renal colic within the emergency department.

DETAILED DESCRIPTION:
Renal colic, an intensely painful condition, is a common presenting complaint to the emergency department. Parenteral opioids, nonsteroidal anti-inflammatory drugs and acetaminophen are commonly used to provide relief from renal colic. The aim of the present trial was to investigate the analgesic efficacy and safety of Transcutaneous electrical nerve stimulation treatment in patients with renal colic within the emergency department.

Study Design and Setting: A prospective, randomized, double-blind, placebo controlled, single-center, clinical trial will be conducted in emergency department of a tertiary care university hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with renal colic admitted to emergency department.
2. Adult patients who were definitively diagnosed with acute renal colic due to urinary system stones using unenhanced computed abdominopelvic tomography

Exclusion Criteria:

1. Patients below 18 years of age
2. Patients with haemodynamic instability, with fever (temperature=38°C [100.4°F]), with evidence of peritoneal inflammation,
3. Patients using any analgesic within the previous 48 hours of emergency department presentation
4. Patients who declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Reduction of the intensity of pain | 0 minutes, 15 minutes and 30 minutes after taking Transcutaneous Electrical Nerve Stimulation application
  Subjects will complete 100 mm visual analog scales at time zero, 15 and 30 minutes after taking Transcutaneous Electrical Nerve Stimulation application

SECONDARY OUTCOMES:
Adverse events | 30 minutes after
  30 minutes after taking Transcutaneous Electrical Nerve Stimulation application

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, M.D., Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simpson PM, Fouche PF, Thomas RE, Bendall JC. Transcutaneous electrical nerve stimulation for relieving acute pain in the prehospital setting: a systematic review and meta-analysis of randomized-controlled trials. Eur J Emerg Med. 2014 Feb;21(1):10-7. doi: 10.1097/MEJ.0b013e328363c9c1. PMID 23839103